CLINICAL TRIAL: NCT04364841
Title: Effects of Bariatric Surgery on Body Image Level and Sexual Life of Individuals
Brief Title: Body Image and Sexuality After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, EBRU YILDIZ, Principal Investigator, Mersin University
Other Study IDs: Sexuality and obesity
Record Dates: First submitted 2020-04-23; First posted 2020-04-28 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Obesity, Morbid; Sexual Dysfunction, Physiological
Keywords: bariatric surgery; body image; sexuality; obesity
MeSH Terms: conditions — Obesity, Morbid; Sexual Dysfunction, Physiological; Sexuality; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 19 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sexual desire may decrease among obese individuals who feel worthless and therefore there may be behaviors that avoid sexuality. Sexuality, one of the activities of daily life, is an issue that is affected by cultural norms and rules and individuals have difficulties expressing their sexual problems comfortably. In a systematic review which is about the effect of bariatric surgery on sexuality; it was emphasized that bariatric surgery, the most widely used treatment in obesity, has positive effects upon reproductive hormones and sexual functions thanks to weight loss. In light of these information above-mentioned; the study was done to examine the correlation between body perception and sexual life before and after bariatric surgery among obese individuals.

DETAILED DESCRIPTION:
Obese individuals who want to learn healthy life behaviors and wish to acquire and to realize behavioral changes that will help them cope with health problems are in need of training and counseling. In this process, nurses -being in close and continuous contact with individuals- play counselor role as a part of their educator roles. It is stated that nurses need to understand, empathize with and support individuals who suffer from different problems while they play this role. In presence of obesity, which is a psychophysiological condition; nurses should also consider the fact that obese individuals who face bitter criticisms and social exclusion may show low self-esteem and impaired body image due to excessive weight and therefore they should give these individuals opportunities to express their feelings as to how they perceive themselves. The studies in literature that investigated the correlation between body mass index (BMI) and self-esteem and body perception report that obese individuals demonstrate relatively lower self-esteem and body perception as compared to the normal individuals. Psychological and hormonal disorders, impaired body image and chronic diseases that develop with obesity influence sexual life negatively, too. Therefore; sexual desire may decrease among obese individuals who feel worthless and therefore there may be behaviors that avoid sexuality. Sexuality, one of the activities of daily life, is an issue that is affected by cultural norms and rules and individuals have difficulties expressing their sexual problems comfortably.

ELIGIBILITY:
Inclusion Criteria:

* Accepted to join the study,
* Did not have such psychiatric disorders as anxiety, depression and personality disorders
* Were aged between 18 and 65.

Exclusion Criteria:

* Do not accepting to join the study,
* Have such psychiatric disorders as anxiety, depression and personality disorders
* Older from 65, under the age of 18.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of the study was consisted of 33 patients who received obesity diagnosis at General Surgery Unit, Mersin University Hospital and underwent bariatric surgery between 1.6.2017 and 1.12.2018. It was identified that the number of the patients who had bariatric surgery at the hospital between 30.11.2016 and 30.5.2017 was 33. During the sampling phase, at least 27 of the 33 patients who volunteered to join the study and met inclusion and exclusion criteria were targeted between 01.06.2017 and 01.12.2018 when Data Collection Forms were distributed according to the statistical calculations in which 20% loss of the population was predicted. However, the whole population was achieved.
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Obese individuals' Descriptive Characteristics and Findings Related to the Disease as assessed by "Information Request Form". | 1 day
  At the first stage of the research, by the obese individuals "Information Request Form" is filled in to specify socio-demographic characteristics.
Obese individuals' Body Perception as assessed by "Body Perception Scale" at the pre-operation period | 1 day
  "Body Perception Scale" filled in to determine how satisfied they were the various parts of their bodies and various body functions at the pre-operation period by the obese individuals.
  The scale includes 40 items and each item refers to an organ or a limb (arm, leg, face, etc.) or a function (sexual activity level). Each item score ranges from 1 to 5 by marking "I do not like at all", "I do not like", "I am uncertain", "I like", "I like a lot". Total score ranges from 40 to 200. High scores indicate high level of satisfaction. Cutoff score of the scale was 135 and scores lower than 135 (≥135) indicate lower body perception.
Obese individuals' sexual functions respective of sexual orientation as assessed by "Arizona Sexual Experiences Scale " at the pre-operation period | 1 day
  The "Arizona Sexual Experiences Scale" was filled in to measure sexual functions related to sexual orientation and the relationship with partners at the pre-operation period by the obese individuals.
  Scores for each question range from 1 to 6 and total score ranges from 5 to 30. Lower scores indicate strong, easy and satisfactory sexual response while higher scores indicate presence of sexual dysfunctions. According to Soykan, a score ≥11 is a cutoff score for sexual dysfunction.

SECONDARY OUTCOMES:
Obese individuals' Body Perception as assessed by "Body Perception Scale" at the post-operation period | 1 day
  "Body Perception Scale" filled in to determine how satisfied they were the various parts of their bodies and various body functions at the post-operation period by the obese individuals.
  The scale includes 40 items and each item refers to an organ or a limb (arm, leg, face, etc.) or a function (sexual activity level). Each item score ranges from 1 to 5 by marking "I do not like at all", "I do not like", "I am uncertain", "I like", "I like a lot". Total score ranges from 40 to 200. High scores indicate high level of satisfaction. Cutoff score of the scale was 135 and scores lower than 135 (≥135) indicate lower body perception.
Obese individuals' sexual functions respective of sexual orientation as assessed by "Arizona Sexual Experiences Scale " at the post-operation period | 1 day
  The "Arizona Sexual Experiences Scale" was filled in to measure sexual functions related to sexual orientation and the relationship with partners at the post-operation period by the obese individuals.
  Scores for each question range from 1 to 6 and total score ranges from 5 to 30. Lower scores indicate strong, easy and satisfactory sexual response while higher scores indicate presence of sexual dysfunctions. According to Soykan, a score ≥11 is a cutoff score for sexual dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University Faculty of Nursing, Mersin, Turkey (Türkiye)

REFERENCES:
- [Background] Kaya H. Patient education in health services and responsibilities of nurse: review. Turkiye Klinikleri Journal of Nursing Sciences. 2009; 1: 19-23.
- [Background] Tedik SE. Healthy life and role of nursing in thecontrol of body weight. TurkishJ ournal of Diabetes and Obesity. 2017; 2: 54-62.
- [Background] Pujols Y, Seal BN, Meston CM. The association between sexual satisfaction and body image in women. J Sex Med. 2010 Feb;7(2 Pt 2):905-16. doi: 10.1111/j.1743-6109.2009.01604.x. Epub 2009 Nov 24. PMID 19968771
- [Background] Hamurcu P, Öner C, Telatar B, Yeşildağ Ş. The impact of obesity on self esteem and body image. Turkish Journal of Family Practice. 2015; 19: 122-128.
- [Background] Wallwiener S, Strohmaier J, Wallwiener LM, Schonfisch B, Zipfel S, Brucker SY, Rietschel M, Wallwiener CW. Sexual Function Is Correlated With Body Image and Partnership Quality in Female University Students. J Sex Med. 2016 Oct;13(10):1530-8. doi: 10.1016/j.jsxm.2016.07.020. Epub 2016 Aug 23. PMID 27567073
- [Background] Hall AM. Sexuality. In (Chapter 28) : Potter, P. A, Perry, A. G. E., Hall, A. E. & Stockert, P. A. (ed.), (2009). Fundamentals of nursing. Elsevier Mosby. pp: 426-442.